CLINICAL TRIAL: NCT02573272
Title: Impact of Eslicarbazepine Acetate on Lipid Metabolism and Cardiovascular Risk Factors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Andalusian Initiative for Advanced Therapies - Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: FPS-ESL-2105-01
Record Dates: First submitted 2015-09-30; First posted 2015-10-09 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Epileptic patients with AEDs and eslicarbacepine
  Interventions: Drug: eslicarbacepine

INTERVENTIONS:
Drug: eslicarbacepine

SUMMARY:
Knowing the impact that the use of ESL as adjunctive treatment of partial epilepsy has on cardiovascular risk factors measured by biochemical and ultrasound parameters compared with enzyme-inducing AEDs.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* patients definitively diagnosed Focal Epilepsy based on clinical criteria and additional tests.
* patients with stable and identifiable antiepileptic treatment during the last two years.
* patients according to the investigator are able to provide clinical data necessary for the development of the study
* Patients who signed informed consent

Exclusion Criteria:

* Patients who, according to their evolution and demands of clinical practice, their previous treatment has to be changed for this reason breach inclusion criteria and / or attachment to one of the study groups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with focal epilepsy on stable treatment for the last two years
Sampling Method: Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Carotid IMT millimeters | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Torrecardenas, Almería, Almeria, Spain